CLINICAL TRIAL: NCT01397396
Title: Effects of Inspiratory Muscle Training in Patients With Chronic Obstructive Pulmonary Disease - a Randomized Controlled Trial
Brief Title: Effects of Inspiratory Muscle Training in COPD
Acronym: IMTCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Daniel Langer, Dr Daniel Langer, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S52852
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: COPD; Inspiratory Muscle Weakness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Inspiratory Muscle Training (Experimental): Inspiratory Muscle Training
  Interventions: Procedure: Inspiratory Muscle Training
- Sham IMT (Placebo Comparator): Sham Inspiratory Muscle Training
  Interventions: Procedure: Inspiratory Muscle Training

INTERVENTIONS:
Procedure: Inspiratory Muscle Training — Three times daily inspiratory muscle training (2x30 breaths) at an intensity of >50% Pi,max

SUMMARY:
The additional effect of inspiratory muscle training as an adjunct to a general exercise training program in patients with COPD with inspiratory muscle weakness will be studied. The main hypothesis is that inspiratory muscle training combined with an exercise training program improves functional exercise capacity more than an exercise training program without the addition of an inspiratory muscle training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD
* Eligible to participate in a exercise training intervention of 8 weeks
* Pi,max <60cmH2O or <50% of the predicted normal value

Exclusion Criteria:

* Major comorbidities preventing successful participation in an 8 week exercise training intervention

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
6-Minute Walking Distance | Baseline and 8 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rik Gosselink, PT, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Charususin N, Gosselink R, Decramer M, Demeyer H, McConnell A, Saey D, Maltais F, Derom E, Vermeersch S, Heijdra YF, van Helvoort H, Garms L, Schneeberger T, Kenn K, Gloeckl R, Langer D. Randomised controlled trial of adjunctive inspiratory muscle training for patients with COPD. Thorax. 2018 Oct;73(10):942-950. doi: 10.1136/thoraxjnl-2017-211417. Epub 2018 Jun 18. PMID 29914940
- [Derived] Charususin N, Gosselink R, Decramer M, McConnell A, Saey D, Maltais F, Derom E, Vermeersch S, van Helvoort H, Heijdra Y, Klaassen M, Glockl R, Kenn K, Langer D. Inspiratory muscle training protocol for patients with chronic obstructive pulmonary disease (IMTCO study): a multicentre randomised controlled trial. BMJ Open. 2013 Aug 5;3(8):e003101. doi: 10.1136/bmjopen-2013-003101. PMID 23921069